CLINICAL TRIAL: NCT02087878
Title: A Multicenter Study to Collect Samples for Future Evaluation of Biomarkers and Genetic Mutations in Patients Exposed to Adalimumab With Crohn's Disease (CD) or Ulcerative Colitis (UC) Who Developed Hepatosplenic T-Cell Lymphoma (HSTCL)
Brief Title: A Blood and Tissue Sample Collection Study of Patients Who Have Inflammatory Bowel Disease, Who Have Been Treated With Adalimumab and Who Developed Hepatosplenic T-Cell Lymphoma
Acronym: HSTCL
Status: Withdrawn | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: F14-258
Record Dates: First submitted 2014-03-13; First posted 2014-03-14 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Crohn's Disease; Ulcerative Colitis (UC); Hepatosplenic T-Cell Lymphoma
Keywords: Hepatosplenic T-Cell Lymphoma
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 1-10 mL blood (serum) for biomarker samples; separate consent for 1- 4 mL whole blood sample for DNA isolation. Biopsy tissue and Fine Needle Aspirate also collected. Samples will be shipped to a designated storage facility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: To collect and store blood and biopsy samples obtained from CD or UC patients exposed to adalimumab and diagnosed with HSTCL for the purpose of identifying potential biomarkers and genetic mutations in patients who develop HSTCL.

SUMMARY:
To collect and store blood and biopsy samples obtained from CD or UC patients exposed to adalimumab and diagnosed with Hepatosplenic T-cell Lymphoma (HSTCL), for the purpose of identifying potential biomarkers and genetic mutations in patients who have developed HSTCL.

DETAILED DESCRIPTION:
A study to bank samples for future evaluation to identify genetic mutations and other biomarkers that predispose inflammatory bowel disease (IBD) patients to developing Hepatosplenic T-cell Lymphoma (HSTCL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female who has received a single dose of HUMIRA prior to a confirmed diagnosis of HSTCL.
* Confirmed diagnosis of CD or UC as documented by a Gastroenterologist or physician who diagnosed the CD or UC.
* Confirmed diagnosis of HSTCL as determined by a biopsy performed on a specimen taken from the patient.
* Patients 18 years old and older must voluntarily sign and date an IRB/EC approved Informed Consent Form. For patients younger than 18 years old, a parent or legal guardian is required to voluntarily sign and date an IRB/EC approved Informed Consent Form. Pediatric patients will be included in all discussions if possible, in order to obtain their assent.

Exclusion Criteria:

* Male or female who has not received at least a single dose of adalimumab prior to a confirmed diagnosis of HSTCL.
* Unconfirmed diagnosis of HSTCL, CD or UC, respectively.
* The patient or the patient's HCP is unwilling to participate in this study.
* The parents or legal guardians (in the case of patients younger than 18 years of age), who are unable and/or unwilling to consent to the patient's participation in this study.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients of any age with CD or UC in the US with HSTCL who are identified through the Sponsor's adverse event reporting systems and who were exposed to HUMIRA prior to the diagnosis of HSTCL.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Collection of Samples | Up to 6 years
  A study to bank blood and tissue samples for future evaluation to identify genetic mutations and other biomarkers that predispose inflammatory bowel disease (IBD) patients to developing Hepatosplenic T-Cell Lymphoma (HSTCL). Samples will be obtained from patients who have Crohn's Disease or Ulcerative Colitis, who have been treated with adalimumab and diagnosed with HSTCL.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (1):
- AOU Pisana /ID# 208952, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided